CLINICAL TRIAL: NCT01751685
Title: Study of Hyperkyphosis, Exercise and Function-SHEAF
Acronym: sheaf
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P0046955; R01AG041921-05 (NIH)
Record Dates: First submitted 2012-12-03; First posted 2012-12-18 (Estimated); Results first posted 2023-03-07 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Kyphosis
Keywords: kyphosis
MeSH Terms: conditions — Kyphosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Kyphosis-specific spinal exercises (Experimental): Investigator developed the intervention protocol (Kyphosis-specific spinal exercises) of targeted spine exercises during our pilot study based upon the literature and clinical experience.We standardized the protocol with a written script and a video. Each exercise session will be preceded by light aerobic activity, ended with cool-down and stretching the neck, chest and all extremities. All participants will be carefully monitored to ensure that all exercises will be performed slowly, with correct body alignment and technique to minimize risk of injury.
  Interventions: Behavioral: Kyphosis-specific spinal strengthening exercises
- Control (Placebo Comparator): Usual care control group will meet once a month for educational lectures on various topics. At the end of 6 months, each control group participant will get a one-on-one session with the physical therapist who was leading the intervention classes.
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: Kyphosis-specific spinal strengthening exercises — Investigator developed the intervention protocol (Kyphosis-specific spinal strengthening exercises) of targeted spine exercises during our pilot study based upon the literature and clinical experience.We standardized the protocol with a written script and a video. Each exercise session will be preceded by light aerobic activity, ended with cool-down and stretching the neck, chest and all extremities. All participants will be carefully monitored to ensure that all exercises will be performed slowly, with correct body alignment and technique to minimize risk of injury.
  Arms: Kyphosis-specific spinal exercises
Other: Control — monthly educational lectures on various topics
  Arms: Control

SUMMARY:
We propose to conduct a randomized, controlled trial among 100 men and women aged 60 or older with hyperkyphosis to an exercise intervention that includes kyphosis-specific spinal muscle strengthening exercises compared to a usual care control group. The study will be conducted in five waves,with 10 participants in the exercise intervention and 10 participants in the control group in each wave.

DETAILED DESCRIPTION:
The experimental interventions will be provided in small groups meeting three sessions per week for 6 months. At baseline and 6 months after the intervention, we will measure kyphosis, physical function, spine muscle strength and density, and quality of life. We will assess the effect of the intervention on the co-primary outcomes of kyphosis, modified Physical Performance Test (PPT) and gait speed measured as change over 6 months. We will also assess the effect of the intervention on secondary outcomes of physical function and health-related quality of life, measured as change in Timed Up and Go, Timed Loaded Standing, Six-Minute Timed Walk, the Scoliosis Research Society SRS-30, PROMISe Global Health and physical function and PACE questionnaires. Furthermore, we will investigate whether changes in kyphosis, spinal muscle strength and/or density mediate the effect of the intervention on change in physical function. After the 6-month intervention, both groups will continue their usual activity and we will assess the durability of the effects of the intervention at 1-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 years and older, kyphosis angle >= 40 degrees measured by kyphometer, medical approval from study physician and primary care provider to participate in exercise intervention

Exclusion Criteria:

* Gait speed <0.6 meters/sec, inability to rise from a chair with arms crossed at chest, painful vertebral fractures in the past 3 months, 3 or more falls in the past year, advanced disability or end-stage disease, major psychiatric illness, cognitive impairment, alcohol, drug abuse, or narcotic pain medications, uncontrolled hypertension, peripheral neuropathy associated with type I diabetes, chest pain, myocardial infarction, or cardiac surgery within the previous 6 months, diagnosed vestibular or neurologic disorder, total hip or knee replacement or hip fracture within previous 6 months, oral glucocorticoid medications for ≥ 3 months the past year, no active movement in thoracic spine, unable to execute exercise safety tests, failure to comply with run-in procedures: poor attendance, or use of actigraph, non-English speaking

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2013-02-01 (Actual); Primary Completion 2016-07-01 (Actual); Study Completion 2019-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wendy B Katzman, DPTSc, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF, San Francisco, California, United States

REFERENCES:
- [Background] Katzman WB, Vittinghoff E, Kado DM, Schafer AL, Wong SS, Gladin A, Lane NE. Study of Hyperkyphosis, Exercise and Function (SHEAF) Protocol of a Randomized Controlled Trial of Multimodal Spine-Strengthening Exercise in Older Adults With Hyperkyphosis. Phys Ther. 2016 Mar;96(3):371-81. doi: 10.2522/ptj.20150171. Epub 2015 Aug 6. PMID 26251480
- [Result] Katzman WB, Vittinghoff E, Lin F, Schafer A, Long RK, Wong S, Gladin A, Fan B, Allaire B, Kado DM, Lane NE. Targeted spine strengthening exercise and posture training program to reduce hyperkyphosis in older adults: results from the study of hyperkyphosis, exercise, and function (SHEAF) randomized controlled trial. Osteoporos Int. 2017 Oct;28(10):2831-2841. doi: 10.1007/s00198-017-4109-x. Epub 2017 Jul 8. PMID 28689306

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Speaks English, age ≥60 years, kyphosis angle ≥40° by the Debrunner kyphometer measured at the screening visit, and ability to walk one block without the use of an assistive device, climb one flight of stairs independently, and rise from a chair without the use of one's arms. Participants were excluded for inability to straighten the thoracic spine at least 5°, cognitive impairment, inability to pass safety tests in screening or any disorder or disease likely to interfere with safe participation
Period: 6-mo Followup
Arm/Group | Kyphosis-specific Spinal Exercises | Control
Started | 51 | 48
Completed | 48 | 45
Not Completed | 3 | 3
Not completed — Missed study visit | 1 | 0
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Lost to Follow-up | 0 | 1
Period: 12-mo Followup
Arm/Group | Kyphosis-specific Spinal Exercises | Control
Started | 48 | 45
Completed | 43 | 45
Not Completed | 5 | 0
Not completed — Lost to Follow-up | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Kyphosis-specific Spinal Exercises | Control | Total
Number analyzed (Participants) | 51 | 48 | 99
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 51 | 48 | 99
Age, Continuous [Mean (Full Range); unit: years] | 71.0 [64.5 to 77.5] | 70.2 [64.5 to 75.9] | 70.6 [64.5 to 75.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 36 | 71
  Male | 16 | 12 | 28
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 51 | 48 | 99

OUTCOME MEASURES:

1. Primary Outcome: Change in Cobb Angle of Kyphosis
Description: The primary outcome is change in kyphosis from baseline to 6 months, measured using the gold standard Cobb angle of kyphosis derived from standing lateral spine radiographs and a standardized protocol for thoracic kyphosis (T4-T12). The study team performed exploratory analyses using the centroid method for measuring Cobb angle from lateral spine radiograph and the Debrunner kyphometer external measurement of kyphosis. Participants stood barefoot with knees straight and arms supported at 90° of flexion; they were instructed to hold full inhalation for the duration of the scan. Measurements were made by a trained radiologist (BF) who read the radiographs paired by participant but blinded to group allocation. A greater Cobb angle indicates more kyphosis severity.
Time Frame: Baseline and 6 months
Measure: Mean (95% Confidence Interval); unit: Degrees
Arm/Group | Kyphosis-specific Spinal Exercises | Control
Number analyzed (Participants) | 51 | 48
Degrees | -3.3 [-4.9 to -1.7] | -0.3 [-1.9 to 1.2]

2. Secondary Outcome: Change in Modified Physical Performance Test (PPT)
Description: Modified Physical Performance Test (PPT) is a composite measure of physical function in aging adults: 50ft [15.2-m] floor walk, putting on and removing a laboratory coat, picking up a penny from the floor, standing up 5 times from a 40.6cm-high [16in-high] chair without the use of arms, lifting a 7-lb book to a shelf, climbing one flight of stairs, and standing with feet together) and 2 additional untimed tasks (climbing up and down 4 flights of stairs and performing a 360° turn).
  The test involves 9 functional items, 4 points per item; the range is 0-36 points, and higher values represent a higher physical performance.
Time Frame: Baseline and 6 months
Measure: Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Kyphosis-specific Spinal Exercises | Control
Number analyzed (Participants) | 51 | 48
Score on a scale | 0.3 [-0.2 to 0.8] | 0.8 [0.3 to 1.3]

3. Other Pre Specified Outcome: Effect of Exercise Intervention on Kyphosis
Description: Investigators will measure change in Cobb angle on lateral spine radiograph.
Time Frame: 1 year post baseline
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Effect of Exercise Intervention on Secondary Measure of Physical Function
Description: Investigators will measure change in physical function with Modified Physical Performance Test (PPT), gait speed, Timed Up and Go, Timed Loaded Standing, 6 minute walk and spinal extensor muscle strength.
Time Frame: 1-year post baseline
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Effect of Exercise Intervention on Health Related Quality of Life (HRQOL)
Description: Investigators will measure change in HRQOL with the Scoliosis Research Society SRS-30 (self image domain) and PROMIS Physical Function and Global Health questionnaires.
Time Frame: 6 month post baseline
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Effect of Exercise Intervention on Health Related Quality of Life (HRQOL)
Description: as for outcome 5
Time Frame: 1 year post baseline
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Effect of Exercise Intervention on Muscle Strength
Description: Investigators will measure change in spinal muscle strength as measured with a Biodex computerized dynamometer, and spinal muscle density as measured with quantitative computed tomography.
Time Frame: 6 month post baseline
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year
Description: Participants are asked to report adverse events to the study staff. Serious adverse events (death, life-threatening adverse experiences, related inpatient hospitalization) will be reported to the University of California, San Francisco Committee on Human Subjects Research in 5 days.
Arm/Group | Kyphosis-specific Spinal Exercises | Control
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/48
Other Adverse Events (participants affected / at risk) | 37/51 | 17/48
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Kyphosis-specific Spinal Exercises (N=51) | Control (N=48)
Falls (Musculoskeletal and connective tissue disorders) | 13 (13) | 8 (8)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 30 (30) | 12 (12)

LIMITATIONS AND CAVEATS:
A healthy community-based group of adults ≥60 years of age were recruited and individuals with comorbidities that could interfere with safe participation in a group exercise class were excluded. Blinding the participants and the instructors providing the intervention is not possible. Although such blinding is not uncommon in exercise trials, it was ensured that the investigators measuring kyphosis and performing the physical function testing are blinded to group allocation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2012-08-03): https://cdn.clinicaltrials.gov/large-docs/85/NCT01751685/Prot_SAP_ICF_000.pdf